CLINICAL TRIAL: NCT04834349
Title: A Phase II Study of Reirradiation With NBTXR3 in Patients With Inoperable Locoregional Recurrent Head and Neck Squamous Cell Carcinoma
Brief Title: Re-irradiation With NBTXR3 in Combination With Pembrolizumab for the Treatment of Inoperable Locoregional Recurrent Head and Neck Squamous Cell Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants were enrolled
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0354; NCI-2021-00123 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0354 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-03-05; First posted 2021-04-08 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Head and Neck Squamous Cell Carcinoma; Unresectable Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy, Intensity-Modulated; pembrolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (NBTXR3, SBRT, pembrolizumab) (Experimental): Patients receive NBTXR3 IT on day 1. Patients then undergo SBRT QOD on days 15-29. Beginning the first day of radiation therapy, patients also receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Hafnium Oxide-containing Nanoparticles NBTXR3; Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy
- Cohort II (NBTXR3, IMRT/IMPT, pembrolizumab) (Experimental): Patients receive NBTXR3 IT on day 1. Patients then undergo IMRT/IMPT QD on days 15-50. Beginning the first day of radiation therapy, patients also receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Hafnium Oxide-containing Nanoparticles NBTXR3; Procedure: Intensity-Modulated Proton Therapy; Radiation: Intensity-Modulated Radiation Therapy; Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Hafnium Oxide-containing Nanoparticles NBTXR3 — Given IT
  Other Names: NBTXR3
Procedure: Intensity-Modulated Proton Therapy — Undergo IMPT
  Other Names: IMPT
  Arms: Cohort II (NBTXR3, IMRT/IMPT, pembrolizumab)
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
  Arms: Cohort II (NBTXR3, IMRT/IMPT, pembrolizumab)
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Cohort I (NBTXR3, SBRT, pembrolizumab)

SUMMARY:
This phase II trial studies the effect of re-irradiation with NBTXR3 in combination with pembrolizumab in treating patients with head and neck squamous cell cancer that cannot be removed by surgery (inoperable) and has come back (recurrent). NBTXR3 is a drug that is designed to improve the effectiveness (how well something works) of radiation therapy. The drug is injected into a tumor and activated (turned on) by radiation. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Radiation therapy, such as intensity modulated radiation therapy or intensity modulated proton therapy, uses high energy to kill tumor cells and shrink tumors. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving NBTXR3 activated by radiation together with pembrolizumab may help to control head and neck squamous cell cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate progression free survival (PFS) and early clinical benefit in patients treated with hafnium oxide-containing nanoparticles NBTXR3 (NBTXR3) activated by stereotactic body radiation therapy (SBRT) reirradiation, with concurrent pembrolizumab.

II. To assess the safety profile and estimate early clinical benefit of NBXTR3 activated by dose reduction intensity modulated radiation therapy (IMRT) or intensity modulated proton therapy (IMPT) reirradiation with concurrent pembrolizumab, in subjects with locoregional recurrent head and neck squamous cell carcinoma (HNSCC) not eligible for SBRT.

SECONDARY OBJECTIVES:

I. To evaluate tumor response after NBTXR3 activated by SBRT reirradiation with concurrent pembrolizumab.

II. To evaluate tumor response after NBTXR3 activated by dose reduction IMRT/IMPT reirradiation with concurrent pembrolizumab.

III. To evaluate the safety profile of NBTXR3 activated by SBRT reirradiation with concurrent pembrolizumab.

IV. To evaluate time-to-event outcomes of NBTXR3 activated by SBRT reirradiation with concurrent pembrolizumab.

V. To evaluate time-to-event outcomes of NBTXR3 activated by dose reduction IMRT/IMPT reirradiation with concurrent pembrolizumab.

EXPLORATORY OBJECTIVES:

I. To evaluate lymphedema/fibrosis & dysphagia-related toxicities and functional outcomes of treatment with NBTXR3 activated by SBRT or IMRT or IMPT reirradiation and concurrent pembrolizumab.

II. To assess functional and patient reported outcomes (PRO) of treatment with NBTXR3 activated by SBRT or IMRT or IMPT reirradiation and concurrent pembrolizumab.

III. To associate radiomic measurements with outcomes of treatment with NBTXR3 activated by SBRT or IMRT or IMPT reirradiation and concurrent pembrolizumab.

IV. To evaluate biomarkers of response in subjects treated with NBTXR3 activated by SBRT or IMRT or IMPT reirradiation and concurrent pembrolizumab.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients receive NBTXR3 intratumorally (IT) on day 1. Patients then undergo SBRT every other day (QOD) on days 15-29. Beginning the first day of radiation therapy, patients also receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.

COHORT II: Patients receive NBTXR3 IT on day 1. Patients then undergo IMRT/IMPT every day (QD) on days 15-50. Beginning the first day of radiation therapy, patients also receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven locoregional recurrent squamous cell carcinoma of the head and neck, or second primary HNSCC
* Previous documented receipt of at least 30 Gy and up to 70 Gy of radiation for HNSCC with overlapping fields based on actual dose, prescription percentage

  * 30 Gy for conventional fractionation
  * 15 Gy for hypofractionation
  * 10 Gy for single fraction
* Time interval from prior radiotherapy to NBTXR3 injection (day 1) of at least 6 months
* Not eligible (unresectable) or poor candidate or patient refusal of surgery for HNSCC recurrence
* Amenable to undergo the image guided intratumoral/intranodal injection of NBTXR3 by Interventional Radiologist or ear, nose, and throat (ENT) surgeon, as per investigator or treating physician
* The target lesion(s) in the head and neck should be measurable as per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 on cross sectional imaging and repeated measurements at the same anatomical location should be achievable

  * Up to 3 target lesions may be injected with NBTXR3 and radiated, including the primary tumor and involved lymph node(s)

    * SBRT cohort: =< 60 cm^3 per site, total volume =< 120 cm^3
    * IMRT/IMPT cohort: =< 120 cm^3 per site, total volume =< 200 cm^3
  * Nodal target lesions must be >= 15mm (short axis) based on computed tomography (CT) (slice thickness of 5 mm or less) or magnetic resonance imaging (MRI)
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelet count >= 100,000/mm^3
* Leukocytes >= 1500/mm^3
* Creatinine =< 1.5 x upper limit of normal (ULN)
* Calculated (Calc.) creatinine clearance > 30 mL/min
* Total bilirubin =< 1.5 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
* Serum albumin > 3.5 g/L
* Negative urine or serum pregnancy test =< 7 days prior to NBTXR3 injection in all women of child-bearing potential (WOCBP). WOCBP must agree to follow instructions for method(s) of contraception for the duration the entire study period and 6 months after the last dose of pembrolizumab treatment. Local laws and regulations may require use of alternative and/or additional contraception methods. WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements but should still undergo pregnancy testing
* Signed informed consent form (ICF) indicating that participant understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

* Locoregional relapse with skin ulceration
* Head and neck carcinoma with radiographic evidence of metastasis at screening
* Surgery to the head and neck

  * Excluding diagnostic biopsy
* History of severe immune-related adverse events observed with previous immunotherapy (anti-PD-1/L1) or known sensitivity (grade >= 3) to any excipients
* Has received any approved or investigational anti-neoplastic agent within 4 weeks prior to NBTXR3 injection

  * Except anti-PD-1 therapy, which will not require a washout window
  * Note: a reduced washout window may be considered for therapies with short half-lives (i.e., kinase inhibitors) after discussion with Nanobiotix and investigator
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs)

  * Replacement therapy (i.e., thyroxine, insulin, or physiologic corticosteroid replacement [=< 10 mg prednisone] therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has not recovered from adverse events (AEs) due to previous anti-neoplastic or immune-oncology therapy and/or interventions (including radiation) to =< grade 1

  * Participants with alopecia and =< grade 2 neuropathy may be eligible
* Any live-virus vaccine therapy used for prevention of infectious diseases administered within 4 weeks prior to NBTXR3 injection

  * Except killed-virus Influenza vaccine
  * Exception of other vaccines (e.g. pneumonia) is at the discretion of the treating physician after conducting a personalized risk assessment on a case by case basis
* Prior allogenic stem cell transplantation or organ allograft
* Known contraindication to iodine-based or gadolinium-based IV contrast
* Active malignancy, in addition to head and neck carcinoma, with the exception of basal cell carcinoma of the skin definitively treated and relapse free within at least 1 year since diagnosis or low risk prostate cancer
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, renal failure, cardiac arrhythmia, or psychiatric illness that would limit compliance with treatment
* Known active, uncontrolled (high viral load) human immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection
* Female patients who are pregnant or breastfeeding
* Women of child-bearing potential and their male partners who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and up to 6 months, for females, and 220 days for males after the last dose of pembrolizumab

  * Acceptable methods of contraception are those that, alone or in combination, result in a failure rate of < 1% per year when used consistently and correctly
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From NBTXR3 injection to local or regional recurrence, local or regional progression, distant (outside the head and neck region) progression, or death from any cause, whichever occurs first, assessed up to 5 years
  Will be estimated using the method of Kaplan-Meier. Median times and 95% confidence intervals will also be estimated.
Early clinical benefit activated by SBRT reirradiation | At 6-months post radiation therapy (RT)
  Defined as radiographic evidence of complete response (CR), partial response (PR) or stable disease (SD)
Incidence of acute adverse events activated by dose reduction IMRT or IMPT reirradiation | Up to 90 days post RT
  Will assess treatment related acute and late onset toxicities defined as any grade >= 3 adverse event (AE), excluding dermatitis and mucositis as per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Incidence of late adverse events activated by dose reduction IMRT or IMPT reirradiation | From 90 days post RT to end of study (up to 5 years) From 90 days post RT to end of study (up to 5 years)
  Will assess treatment related acute and late onset toxicities defined as any grade >= 3 AE, excluding dermatitis and mucositis as per NCI CTCAE v 5.0.
Incidence of late adverse events activated by SBRT reirradiation | From 90 days post RT to end of study (up to 5 years)
  Will assess treatment related acute and late onset toxicities defined as any grade >= 3 AE, excluding dermatitis and mucositis as per NCI CTCAE v 5.0.

SECONDARY OUTCOMES:
Objective response rate | Up to 5 years post treatment
  Defined as complete or partial response per RECIST v1.1 in the target lesion(s), which are those injected with NBTXR3 and irradiated.
  All other malignant lesions that have not received NBTXR3 injection will be evaluated as per RECIST v1.1, i.e. as measurable or non-measurable lesions (according to their characteristics) and included for the determination of best objective response.
Overall response | Up to 5 years post treatment
  Evaluated as per RECIST v1.1
Incidence of acute adverse events activated by SBRT reirradiation | Up to 90 days post RT
  Will assess treatment related acute and late onset toxicities defined as any grade >= 3 AE, excluding dermatitis and mucositis as per NCI CTCAE v 5.0.
Local PFS | From NBTXR3 injection to the radiographic and/or histological confirmation of local (within 2 cm of the high-dose reirradiation treatment volume [PTV]) disease recurrence, local progression, or death from any cause, assessed up to 5 years
  Will be estimated using the method of Kaplan-Meier. Median times and 95% confidence intervals will also be estimated.
Regional PFS | From NBTXR3 injection to the radiographic and/or histological confirmation of regional disease recurrence, regional progression, or death from any cause, whichever occurs first, assessed up to 5 years
  Will be estimated using the method of Kaplan-Meier. Median times and 95% confidence intervals will also be estimated.
Distant PFS | From NBTXR3 injection to the radiographic and/or histological confirmation of a new lesion outside the head and neck region, or death from any cause, whichever occurs first, assessed up to 5 years
  Will be estimated using the method of Kaplan-Meier. Median times and 95% confidence intervals will also be estimated.
Overall survival | From NBTXR3 injection to death from any cause or EoS, whichever occurs first, assessed up to 5 years
  Will be estimated using the method of Kaplan-Meier. Median times and 95% confidence intervals will also be estimated.

OTHER OUTCOMES:
Evaluation of the clinical-grading of lymphedema/fibrosis | Up to 5 years post treatment
  Evaluation of the clinical-grading of lymphedema/fibrosis according to the Head and Neck-Lymphedema Fibrosis (HN-LEF)
  Lymphedema/Fibrosis Grading: Clinician-grading of lymphedema/fibrosis will be conducted according to the published Head and Neck-Lymphedema Fibrosis (HN-LEF) per physical examination of the patient. Clinical grading is a brief assessment that can be completed in < 5 minutes.
Evaluation of the clinical-grading of lymphedema/fibrosis | Up to 5 years post treatment
  Evaluation of the clinical-grading of lymphedema/fibrosis according Cervical range of motion (CROM) per physical examination of patient.
  Cervical range of motion (CROM): A goniometer will measure CROM (degrees) to assess active cervical spine ROM. Five core CROM measures will be collected, including cervical extension, sagittal plane at rest, lateral flexion (left/right), coronal plane at rest, and lateral rotation (left/right). The primary CROM measure of interest is cervical extension. Cervical extension measures are highly reliable (ICC=.90). Average extension measures in healthy adults aged 60 to 69 range from 57 degrees in males (SD: 10.5) to 65 degrees in females (SD: 13.3). Cervical extension measures decrease by approximately 5 degrees for each decade of life[41].
Evaluation of the clinical-grading of lymphedema/fibrosis | Up to 5 years post treatment
  Evaluation of the clinical-grading of lymphedema/fibrosis according to the Lymphedema Symptom Intensity and Distress Survey - Head and Neck (LSIDS-H&N).
  Lymphedema Symptom Intensity and Distress Survey - Head and Neck (LSIDS-H&N)25 is a 64-item instrument designed to assess lymphedema symptoms in head and neck cancer patients. Survey items were selected to address six domains (head and neck-specific functioning, systemic symptoms, psychosocial issues, altered sensation symptoms, neck-shoulder musculoskeletal/skin symptoms, and miscellaneous symptoms) identified by an expert panel. Preliminary testing of LSIDS-H&N demonstrated both feasibility and readability.
Patient reports outcomes | Up to 5 years post treatment
  Questionnaires measuring the patients' views of their health status
Biomarkers of response | Up to 5 years post treatment
  Multiplex IHC (mIHC) analysis of tumor microenvironment (i.e. CD8, PD-L1, PD1, CD3, CD68, FoxP3, etc.) in biopsies
  Flow cytometry analysis (cell counts) of the immune cell biomarkers in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Phan, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org